CLINICAL TRIAL: NCT07390864
Title: Intramyometrial Ergometrine Injection Versus Intramyometrial Carbetocin Injection to Decrease Blood Loss During and After Abdominal Myomectomy: A Randomized Clinical Trial
Brief Title: Ergometrine Versus Carbetocin to Decrease Blood Loss in Myomectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, Assistant lecturer of obstetrics and gynecology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Fayoum-MD-2024
Record Dates: First submitted 2026-01-17; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Myoma;Uterus
Keywords: Ergometrine; Carbetocin; Blood Loss; Abdominal Myomectomy
MeSH Terms: conditions — Myofibroma; Hemorrhage | interventions — Methylergonovine; Ergonovine; carbetocin

STUDY DESIGN:
Intervention Model Description: This study is designed as a parallel-group interventional clinical trial. Eligible participants undergoing abdominal myomectomy will be randomly assigned in a 1:1 allocation ratio to one of two intervention arms. Each participant will receive only one study intervention, and no crossover between treatment arms will occur during the study period.
  The parallel design allows for a direct comparison between intramyometrial methylergometrine and intramyometrial carbetocin, with both interventions administered at the same intraoperative time point and under identical surgical conditions. This model minimizes contamination between treatment arms and ensures that observed differences in blood loss and perioperative outcomes can be attributed to the assigned uterotonic agent.
  Randomization will be performed using a computer-generated randomization sequence, and allocation concealment will be maintained through the use of sequentially numbered opaque sealed envelopes. Double blinding will be i
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intramyometrial Ergometrine Injection (Active Comparator): Participants receive intramyometrial injection of methylergometrine maleate diluted in saline and administered circumferentially around the myoma before uterine incision during abdominal myomectomy.
  Interventions: Drug: Methylergometrine (Intramyometrial Injection)
- Intramyometrial Carbetocin Injection (Experimental): Participants receive intramyometrial injection of carbetocin diluted in saline and administered circumferentially around the myoma before uterine incision during abdominal myomectomy.
  Interventions: Drug: Carbetocin (Intramyometrial Injection)

INTERVENTIONS:
Drug: Methylergometrine (Intramyometrial Injection) — Methylergometrine maleate is administered as an intramyometrial injection diluted in normal saline and injected circumferentially around the myoma before uterine incision during abdominal myomectomy to induce sustained uterine contraction and reduce surgical blood loss.
  Other Names: Methylergometrine maleate; Ergometrine; Methergine
  Arms: Intramyometrial Ergometrine Injection
Drug: Carbetocin (Intramyometrial Injection) — Carbetocin is administered as an intramyometrial injection diluted in normal saline and injected circumferentially around the myoma before uterine incision during abdominal myomectomy to promote sustained uterine contraction and reduce intraoperative and postoperative blood loss.
  Other Names: Carbetocin; Long-acting oxytocin analogue
  Arms: Intramyometrial Carbetocin Injection

SUMMARY:
The goal of this randomized clinical trial is to determine whether intramyometrial ergometrine injection or intramyometrial carbetocin injection is more effective in reducing blood loss during and after abdominal myomectomy in women undergoing surgery for symptomatic uterine fibroids.

The main questions it aims to answer are:

Does intramyometrial ergometrine reduce intraoperative and postoperative blood loss during abdominal myomectomy?

Does intramyometrial carbetocin reduce intraoperative and postoperative blood loss during abdominal myomectomy?

Is there a difference between the two drugs in the need for blood transfusion and postoperative hemoglobin drop?

Researchers will compare intramyometrial ergometrine injection with intramyometrial carbetocin injection to see which intervention is more effective in controlling surgical bleeding and improving surgical outcomes.

Participants will:

Undergo abdominal myomectomy for uterine fibroids

Receive either intramyometrial ergometrine or intramyometrial carbetocin during surgery

Be monitored for intraoperative blood loss, postoperative blood loss, hemoglobin changes, and need for blood transfusion

DETAILED DESCRIPTION:
Uterine leiomyomas are the most common benign tumors of the female reproductive tract and frequently require surgical management when symptomatic. Abdominal myomectomy remains the standard fertility-preserving surgical option for women with large or multiple intramyometrial fibroids. However, excessive intraoperative and postoperative blood loss continues to be a major challenge during myomectomy and is associated with increased morbidity, blood transfusion requirements, prolonged hospitalization, and delayed recovery.

Several pharmacological and surgical strategies have been investigated to minimize blood loss during myomectomy, including mechanical tourniquets, vasoconstrictors, uterine artery occlusion, and uterotonic agents. Among uterotonics, methylergometrine maleate and carbetocin are well-established agents that induce sustained uterine contractions and may reduce bleeding by compressing uterine vasculature. Methylergometrine, an ergot alkaloid, has long been used in obstetric hemorrhage, while carbetocin, a long-acting oxytocin analogue, offers prolonged uterotonic activity with a favorable pharmacokinetic profile. Despite their individual use, comparative data on their intramyometrial administration during abdominal myomectomy remain limited.

This prospective, double-blind, randomized comparative clinical trial is designed to evaluate and compare the effectiveness of intramyometrial methylergometrine versus intramyometrial carbetocin in reducing blood loss during and after abdominal myomectomy. The study will be conducted at Fayoum University maternity hospitals over an anticipated period of 20 months. To minimize bias, all procedures will be performed by the same surgical team following a standardized operative technique.

Participants will be randomly allocated to one of two intervention arms. In the first arm, methylergometrine maleate diluted in saline will be injected intramyometrially around the myoma before uterine incision. In the second arm, carbetocin diluted in saline will be administered in the same intramyometrial manner. The injections will be given circumferentially around the myoma, approximately 1-2 cm from its margins, and repeated as needed according to the number of myomas. Allocation concealment will be ensured using sequentially numbered opaque sealed envelopes, and double blinding will be maintained by coding the study drugs, with the allocation key retained by a designated supervisor until study completion.

A standardized abdominal myomectomy technique will be used in all cases, including Pfannenstiel incision, careful enucleation of myomas, meticulous hemostasis, layered uterine closure, and routine use of intraperitoneal drainage. Intraoperative blood loss will be quantified using a gravimetric method combined with suction measurements, while postoperative blood loss will be assessed via drain output. Perioperative monitoring will include vital signs, laboratory investigations, and clinical assessment for adverse events.

Safety monitoring will focus on drug-related side effects, hemodynamic changes, thromboembolic manifestations, and postoperative complications. The need for intraoperative or postoperative blood transfusion will be determined according to predefined clinical and laboratory criteria. Participants will be followed postoperatively until discharge and reassessed during early follow-up to ensure recovery and detect delayed complications.

The findings of this study are expected to provide evidence-based guidance on the optimal intramyometrial uterotonic agent for reducing blood loss during abdominal myomectomy, thereby improving surgical safety and patient outcomes in gynecologic practice.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 25 to 48 years
* Body mass index (BMI) < 35 kg/m²
* Symptomatic uterine fibroids requiring surgical management (e.g., abnormal uterine bleeding, pelvic pain, or pressure symptoms)
* Intramyometrial uterine myomas classified as FIGO types 3 to 6, diagnosed by transvaginal ultrasonography or magnetic resonance imaging
* Maximum diameter of the largest myoma ≤ 20 cm
* Eligible for and scheduled to undergo abdominal myomectomy
* Able and willing to provide written informed consent

Exclusion Criteria:

* FIGO type 0, 1, 2, 7, or 8 myomas (intracavitary, submucosal, pedunculated subserosal, cervical, or adnexal)
* History of pelvic inflammatory disease, peritonitis, or significant abdominal or pelvic infection
* History of prior uterine surgery
* Use of hormonal treatment within 3 months prior to enrollment
* Contraindication to methylergometrine or carbetocin, including:
* Known drug allergy
* Hypertension
* Cardiac or pulmonary disease
* Chronic endocrine or metabolic disease (e.g., diabetes mellitus)
* Renal or hepatic impairment
* High risk of bleeding, including:
* Known bleeding disorders
* Current use of antiplatelet or anticoagulant therapy
* Preoperative anemia (hemoglobin < 10 g/dL)
* BMI ≥ 35 kg/m²
* Intraoperative conversion from myomectomy to hysterectomy

Ages: 25 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is open to participants who self-identify as female, as the intervention is performed in individuals with a uterus undergoing abdominal myomectomy for uterine fibroids.
Enrollment: 40 (Estimated)
Dates: Start 2026-01-18 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Estimated Intraoperative and Postoperative Blood Loss | From the start of surgery until removal of the intraperitoneal drain (up to 48 hours postoperatively)
  Total blood loss will be assessed as the sum of intraoperative and postoperative blood loss during abdominal myomectomy. Intraoperative blood loss will be estimated using a gravimetric method by weighing surgical swabs and measuring blood volume collected in suction devices. Postoperative blood loss will be measured as the volume collected in the intraperitoneal suction drain.

SECONDARY OUTCOMES:
Need for Blood Transfusion | Intraoperative period and through postoperative day 2 (up to 48 hours after surgery)
  The proportion of participants requiring intraoperative or postoperative blood transfusion will be recorded based on clinical condition and predefined laboratory criteria.
Change in Postoperative Hemoglobin and Hematocrit Levels | Baseline (preoperative) and postoperative day 2 (≈48 hours after surgery)
  Hemoglobin and hematocrit levels will be measured preoperatively and on the second postoperative day to assess perioperative blood loss and the development of postoperative anemia.
Incidence of Drug-Related Side Effects | Time Frame: From drug administration through postoperative day 2 or hospital discharge, whichever occurs first (up to 72 hours)
  The occurrence of adverse effects potentially related to the study drugs, including nausea, vomiting, diarrhea, shivering, headache, and cardiovascular effects, will be monitored and recorded.
Duration of Surgery | During the surgical procedure
  The total operative time will be recorded from skin incision to skin closure to assess surgical efficiency.
Postoperative Febrile Morbidity | From end of surgery through postoperative day 3 (up to 72 hours after surgery)
  The incidence of postoperative fever will be recorded as an indicator of infection or other postoperative complications.
Length of Postoperative Hospital Stay | From date of surgery to hospital discharge (up to 7 days)
  The duration of hospital stay will be measured in days from the date of surgery until discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet determined whether de-identified individual participant data (IPD) will be shared. If sharing is approved, only de-identified IPD necessary to reproduce the primary analyses may be made available to qualified researchers, and results will also be reported in aggregate form in publications.

REFERENCES:
- [Result] Taher A, Farouk D, Mohamed Kotb MM, Ghamry NK, Kholaif K, A Mageed A Allah A, Ali AS, Osman OM, Nabil H, Islam Y, Bakry MS, Islam BA, Alalfy M, Nassar SA, Bosilah AH, Ghanem AA, Ali Rund NM, Refaat R, Abdel Wahed Ali HA, Bakry A, Ashour ASA, Nabil M, Zaki SS. Evaluating efficacy of intravenous carbetocin in reducing blood loss during abdominal myomectomy: a randomized controlled trial. Fertil Steril. 2021 Mar;115(3):793-801. doi: 10.1016/j.fertnstert.2020.09.132. Epub 2021 Jan 16. PMID 33461754
- [Result] Gallos I, Williams H, Price M, Pickering K, Merriel A, Tobias A, Lissauer D, Gee H, Tuncalp O, Gyte G, Moorthy V, Roberts T, Deeks J, Hofmeyr J, Gulmezoglu M, Coomarasamy A. Uterotonic drugs to prevent postpartum haemorrhage: a network meta-analysis. Health Technol Assess. 2019 Feb;23(9):1-356. doi: 10.3310/hta23090. PMID 30821683
- [Result] Spencer SPE, Lowe SA. Ergometrine for postpartum hemorrhage and associated myocardial ischemia: Two case reports and a review of the literature. Clin Case Rep. 2019 Nov 6;7(12):2433-2442. doi: 10.1002/ccr3.2516. eCollection 2019 Dec. PMID 31893076
- [Result] Hickman LC, Kotlyar A, Shue S, Falcone T. Hemostatic Techniques for Myomectomy: An Evidence-Based Approach. J Minim Invasive Gynecol. 2016 May-Jun;23(4):497-504. doi: 10.1016/j.jmig.2016.01.026. Epub 2016 Mar 9. PMID 26855249
- [Result] Kim T, Purdy MP, Kendall-Rauchfuss L, Habermann EB, Bews KA, Glasgow AE, Khan Z. Myomectomy associated blood transfusion risk and morbidity after surgery. Fertil Steril. 2020 Jul;114(1):175-184. doi: 10.1016/j.fertnstert.2020.02.110. Epub 2020 Jun 10. PMID 32532486
- [Result] Donnez J, Taylor HS, Marcellin L, Dolmans MM. Uterine fibroid-related infertility: mechanisms and management. Fertil Steril. 2024 Jul;122(1):31-39. doi: 10.1016/j.fertnstert.2024.02.049. Epub 2024 Mar 5. PMID 38453041
- [Result] Uimari O, Subramaniam KS, Vollenhoven B, Tapmeier TT. Uterine Fibroids (Leiomyomata) and Heavy Menstrual Bleeding. Front Reprod Health. 2022 Mar 4;4:818243. doi: 10.3389/frph.2022.818243. eCollection 2022. PMID 36303616
- [Result] Eltoukhi HM, Modi MN, Weston M, Armstrong AY, Stewart EA. The health disparities of uterine fibroid tumors for African American women: a public health issue. Am J Obstet Gynecol. 2014 Mar;210(3):194-9. doi: 10.1016/j.ajog.2013.08.008. Epub 2013 Aug 11. PMID 23942040
- [Result] Ahmad A, Kumar M, Bhoi NR, Badruddeen, Akhtar J, Khan MI, Ajmal M, Ahmad M. Diagnosis and management of uterine fibroids: current trends and future strategies. J Basic Clin Physiol Pharmacol. 2023 Mar 30;34(3):291-310. doi: 10.1515/jbcpp-2022-0219. eCollection 2023 May 1. PMID 36989026
- [Result] Yang Q, Ciebiera M, Bariani MV, Ali M, Elkafas H, Boyer TG, Al-Hendy A. Comprehensive Review of Uterine Fibroids: Developmental Origin, Pathogenesis, and Treatment. Endocr Rev. 2022 Jul 13;43(4):678-719. doi: 10.1210/endrev/bnab039. PMID 34741454